CLINICAL TRIAL: NCT03549819
Title: Cannabidiol for the Treatment of Anxiety Disorders: An 8-Week Pilot Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Tilray (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBD_ANX
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia
Keywords: Anxiety Disorders; Cannabidiol; Cannabis
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Agoraphobia; Anxiety Disorders; Marijuana Abuse | interventions — Cannabidiol; Oils; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (CBD) Oil Capsules (Experimental): Pure CBD in sunflower lecithin oil, flexibly dosed at 200-800 mg per day
  Interventions: Drug: Cannabidiol (CBD) Oil Capsules
- Sunflower Lecithin Oil in Capsule (Placebo Comparator): 1-4 capsules daily
  Interventions: Drug: Sunflower Lecithin Oil in Capsule

INTERVENTIONS:
Drug: Cannabidiol (CBD) Oil Capsules — 200 mg CBD- titrated as tolerated up to a maximum 2 capsules twice daily (200 mg- 800 mg total dose)
  Start at 1 capsule/day (at bedtime) for one week and be titrated to 1 capsule twice/daily for one week. At the end of Week 2, dose may be titrated to 1 capsule in the morning and 2 capsules at bedtime; then at the end of Week 4, dose may be titrated to 2 capsules twice daily (the maximum of 800 mg/day total dose)
  Arms: Cannabidiol (CBD) Oil Capsules
Drug: Sunflower Lecithin Oil in Capsule — Start at 1 capsule/day (at bedtime) for one week and be titrated to 1 capsule twice/daily for one week. At the end of Week 2, dose may be titrated to 1 capsule in the morning and 2 capsules at bedtime; then at the end of Week 4, dose may be titrated to 2 capsules twice daily (the maximum of 800 mg/day total dose)
  Arms: Sunflower Lecithin Oil in Capsule

SUMMARY:
This proposed study aims to evaluate the efficacy of daily Cannabidiol (CBD) Oil Capsules in treating symptoms of DSM-5 anxiety disorders, using a two-arm, 8-week randomized, placebo-controlled trial in adults aged 21-65 years. The study will also evaluate the relationship between inflammation, anxiety and CBD using biological markers as well as examine the neuro-cognitive effects of CBD treatment.

DETAILED DESCRIPTION:
The study will be a randomized, double-blind, placebo-controlled parallel design comparing the efficacy and safety of flexibly dosed CBD Oil capsules versus placebo for the treatment of adults, aged 21 to 65 years with a primary Diagnostic and Statistical Manual 5 (DSM-5) anxiety disorder: Generalized Anxiety Disorder (GAD), Social Anxiety Disorder (SAD), Panic Disorder (PD), or agoraphobia. A total 50 participants (n=25/cell) who meet the inclusion criteria will be randomized to receive 1 of 2 treatments in a 1:1 ratio: CBD Oil Capsules or matching placebo, with the possibility of dose titration during this 8-week period. The outcomes of this research will make a significant contribution to enhance our current understanding of the effects of cannabis in anxiety disorders.

To be involved in this study, the study doctor will first check that the participant is qualified. This is called screening, and will involve a clinical assessment, physical exam and urine tests. This visit may take up to 3 hours to complete.

If the participant successfully completes screening the participant will start treatment in one of the two assigned treatment groups. Treatment is 8 weeks. Participants will come to the study clinic 6 times during the treatment phase of the study. Each visit will last 1 to 2 hours. Each visit will involve reporting any side effects that the participant may have experienced, completing questionnaires about mood and anxiety symptoms, sleep, overall functioning and alcohol and drug use. Participants will also be assessed by the study doctor. The first and last visits will also involve blood work and completing a number of tasks on the computer, which measure focus, attention and memory.

Each participant will be involved in the study for a maximum of 10 weeks. This includes the screening visit and follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 21-65 years of age with a primary psychiatric diagnosis of either GAD, SAD, PD or agoraphobia as defined by DSM-5 criteria and a HAM-A score of ≥ 22.
2. Physical exam and laboratory findings without clinically significant abnormalities.
3. Participants must agree to abstain from recreational cannabis use for the duration of the study.
4. Concomitant psychotropic medication use will be allowed provided that the dose has been stable for 8 weeks prior to randomization. (including antidepressants, anti-psychotics, anti-convulsants, benzodiazepines, stimulants, mood stabilizers)
5. The ability to comprehend and satisfactorily comply with protocol requirements.
6. Written informed consent given prior to entering the baseline period of the study.

Exclusion Criteria:

1. Current recreational or medicinal use of cannabis within 4 weeks of study initiation.
2. Participants with a lifetime history of cannabis use disorder or other substance use disorders (except tobacco use disorder)will be excluded.
3. Participants with a lifetime history of daily cannabis use will be excluded.
4. Dose changes of concomitant medication will not be permitted during the study period.
5. Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months), or women who are planning on becoming pregnant.
6. Diagnosis of any of the following mental disorders as defined by the DSM-5: a lifetime history of schizophrenia or any other psychosis, mental retardation, organic medical disorders, bipolar disorder. Entry of patients with obsessive compulsive disorder or posttraumatic stress disorder will be permitted if the anxiety disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample.
7. Major depression will be allowed if not severe (Montgomery Asberg Depression Rating Scale-MADRS ≥ 25). Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviours within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
8. Participants with a family history of psychosis will be excluded.
9. Participants who have a history of adverse reactions to cannabis will be excluded.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | Change from baseline to week 8
  The 14-item HAM-A was developed to assess general anxiety symptoms in a clinical population and has proven sensitive to change with treatment. It is a clinician-rated measure and will be administered at each visit by a trained, blinded rater, using the Structured Interview Guide for the HAM-A. It has 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) are summed up to give a total possible score of 0 (not present) to 56 (very severe), where lower scores indicates less anxiety.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | Change from baseline to week 8
  The CGI-S is a clinician-rated instrument used to assess global severity of symptoms. The CGI-S ranges from 1 (normal, not ill) to 7 (among the most severely ill).
Clinical Global Impression - Improvement (CGI-I) | Change from baseline to week 8
  The CGI-I is a clinician-rated instrument used to assess overall improvement of illness. The CGI-I ranges from 1 (very much improved) to 7 (very much worse).
Generalized Anxiety Disorder-7 (GAD-7) | Change from baseline to week 8
  The GAD-7 is a self-reported questionnaire that measures the severity of various signs of GAD. It contains seven items with a 4-point scale (range: 0 to 3). The total possible score is ranged from 0 to 21, with higher scores representing greater severity of GAD.
Liebowitz Social Anxiety Scale- Self Report (LSAS-SR) | Change from baseline to week 8
  The LSAS-SR is a 24 item scale that provides separate scores for fear and avoidance in social and performance situations with higher scores representing increased social anxiety. The LSAS-SR contains three total scores 1) total fear score (0-72), 2) total avoidance score (0-72) and total overall score (0-144).
Panic and Agoraphobia Scale (PAS) | Change from baseline to week 8
  The PAS is a measure of the severity of illness in patients with panic disorder (with or without agoraphobia). It has 13 items with a 5-point scale (range: 0-4). The total possible score is ranged from 0 to 52, with higher scores representing increased severity of illness. It contains 5 sub-scales: panic attacks, agoraphobic avoidance, anticipatory anxiety, disability, and functional avoidance (health concerns).
Quick Inventory of Depressive Symptomology (QIDS) | Change from baseline to week 8
  The QIDS is a self-report measure of depression. It contains 16 items with a 4-point scale (range: 0 to 3) which assess the severity of the nine diagnostic symptom criteria used in the DSM: Sleep disturbance, sad mood, decrease/increase in appetite/weight, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, and psychomotor agitation/retardation. The total possible score is ranged from 0 to 27, with higher scores representing greater severity of depression.
Sheehan Disability Scale (SDS) | Change from baseline to week 8
  The SDS is a 3 question instrument designed to assess functional impairment associated with mental disorders in three domains: work impairment, social impairment, and impairment of family life or home responsibilities. Each sub-scale score ranges from 0 to 10 and a total disability score, calculated as the sum of scores for each question ranges from 0 to 30. Higher scores reflect greater impairment.
World Health Organization Disability Assessment Scale (WHODAS 2.0) | Change from baseline to week 8
  The WHODAS 2.0 is a 36-item self-administered questionnaire that covers 6 domains of functioning, including: Cognition, mobility, self-care, getting along with people, life activities, participation. Each question ranges from 'none' to 'extreme or cannot do'. The scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed to give a total score that ranges from 0 to 144, with higher scores representing a greater degree of functional limitation.
Insomnia Severity Index (ISI) | Change from baseline to week 8
  The ISI has 7 questions with a 5-point score (range: 0 to 4). The total possible score is ranged from 0 to 28, with higher scores reflecting greater severity of sleep difficulty.
Marijuana Craving Questionnaire | Change from baseline to week 8
  The Marijuana Craving Questionnaire is a 47-item self-report instrument that assesses marijuana craving along four dimensions: compulsivity, emotionality, expectancy, and purposefulness. Each item is answered with a 7-point scale from 1 (strongly disagree) to 7 (strongly agree).
Obsessive Compulsive Inventory-Revised (OCI-R) | Change from baseline to week 8
  The OCI-R is a self-report scale for assessing symptoms of Obsessive-Compulsive Disorder (OCD). It consists of 18 questions with a 5-point scale (range: 0 to 4). The possible range of scores is 0 to 72, with higher scores indicating a greater likelihood of the presence of OCD.
PTSD Checklist (PCL-5) | Change from baseline to week 8
  The PCL-5 is a 20 item self-report measure that assesses symptoms of PTSD. Each item is rated on a 5-point scale from 0 (not at all) to 4 (extremely). The possible range of scores is 0 to 80, with higher scores indicating greater severity of PTSD.
Drug Effects Questionnaire (DEQ) | Change from baseline to week 8
  The DEQ assesses the extent to which participants 1) feel any substance effect(s), 2) feel high, 3) like the effects, 4) dislike the effects, and 5) want more of the substance using 100mm Visual Analog Scales.
Marijuana Withdrawal Checklist | Change from baseline to week 8
  The Marijuana Withdrawal Checklist has 22 items that assess mood, behavioural, and physical symptoms associated with marijuana withdrawal. Each item is rated on a 4-point scale from 0 (none) to 3 (severe). A total score is obtained by summing each of the item totals (range 0 to 66). Higher scores indicated more severe symptoms associated with marijuana withdrawal.
Shipley II: Verbal | Baseline
  Measures verbal intelligence quotient (IQ) - crystallized intelligence
Shipley II: Abstraction | Baseline
  Measures abstract intelligence quotient (IQ) - fluid intelligence
Digits Forward Test | Change from baseline to week 8
  Measures attention
Digits Backward Test | Change from baseline to week 8
  Measures working memory
Go/No-Go Test | Change from baseline to week 8
  Measures behavioural inhibition
Monetary Choice Questionnaire | Change from baseline to week 8
  Measures impulsive decision making
Probabilistic Choice Questionnaire | Change from baseline to week 8
  Measures risky decision making
Trails A and B Task | Change from baseline to week 8
  Measures visual attention and switching
Rey Auditory Verbal Learning Test | Change from baseline to week 8
  Measures short-term auditory-verbal memory
Simple Visual Reaction Time Task | Change from baseline to week 8
  Measures reaction time
Sustained Attention to Response Task | Change from baseline to week 8
  Measures sustained attention
Experimental Drug Purchase Task | Week 8
  Measures drug abuse liability
Inflammatory Markers | Change from baseline to week 8
  Serum levels of IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, TNF-α and IFN-γ

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No